CLINICAL TRIAL: NCT06514027
Title: A Multicenter, Open Phase II Clinical Study on the Safety and Efficacy of BEBT-109 Combined With Chemotherapy as First-Line Treatment for Non-Small Cell Lung Cancer Carrying EGFR Exon 20 Insertion Mutations
Brief Title: Study of BEBT-109 in Subjects With Non-Small Cell Lung Cancer Carrying EGFR Exon 20 Insertion Mutations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-109-P04
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: BEBT-109; EGFR exon 20 insertion mutations; Drug combination; First-line treatment; Safety; Efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Injections; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: This study initially sets up two cohorts. In cohort 1, the treatment is BEBT-109 combined with investigator-selected chemotherapy (injectable pemetrexed disodium combined with carboplatin or cisplatin injection). In cohort 2, the treatment is monotherapy with BEBT-109 (BEBT-109 capsule at a dose of 180mg, taken orally once daily). Based on different dosing regimens of BEBT-109 capsules, cohort 1 is divided into three dose groups: A (BEBT-109 capsule at a dose of 180mg, taken orally once daily), B (BEBT-109 capsule at a dose of 120mg, taken orally twice daily), and C (BEBT-109 capsule at a dose of 120mg, taken orally once daily).
  The decision to initiate cohort 2 will be based on the safety and efficacy results from cohort 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose group A of BEBT-109 combined with investigator-selected chemotherapy (Experimental): BEBT-109 Capsules: Administration and Dosage: Oral administration, 180mg; Frequency and Duration of Administration: Once a day,and 21 days as a treatment cycle.
  Pemetrexed Disodium for Injection: Administration and Dosage: Intravenous infusion, 500mg/m^2; Frequency and Duration of Administration: On the first day of each cycle,and 21 days as a treatment cycle.
  Carboplatin Injection: Administration and Dosage: Intravenous infusion, AUC=5 mg/ml.min, with a single dose not exceeding 800 mg; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Cisplatin Injection: Administration and Dosage: Intravenous infusion, 75 mg/m^2; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Interventions: Drug: BEBT-109 Capsules; Drug: Pemetrexed Disodium for Injection; Drug: Carboplatin Injection; Drug: Cisplatin Injection
- Dose group B of BEBT-109 combined with investigator-selected chemotherapy (Experimental): BEBT-109 Capsules: Administration and Dosage: Oral administration, 120mg; Frequency and Duration of Administration: Twice a day,and 21 days as a treatment cycle.
  Pemetrexed Disodium for Injection: Administration and Dosage: Intravenous infusion, 500mg/m^2; Frequency and Duration of Administration: On the first day of each cycle,and 21 days as a treatment cycle.
  Carboplatin Injection: Administration and Dosage: Intravenous infusion, AUC=5 mg/ml.min, with a single dose not exceeding 800 mg; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Cisplatin Injection: Administration and Dosage: Intravenous infusion, 75 mg/m^2; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Interventions: Drug: BEBT-109 Capsules; Drug: Pemetrexed Disodium for Injection; Drug: Carboplatin Injection; Drug: Cisplatin Injection
- Dose group C of BEBT-109 combined with investigator-selected chemotherapy (Experimental): BEBT-109 Capsules: Administration and Dosage: Oral administration, 120mg; Frequency and Duration of Administration: Once a day,and 21 days as a treatment cycle.
  Pemetrexed Disodium for Injection: Administration and Dosage: Intravenous infusion, 500mg/m^2; Frequency and Duration of Administration: On the first day of each cycle,and 21 days as a treatment cycle.
  Carboplatin Injection: Administration and Dosage: Intravenous infusion, AUC=5 mg/ml.min, with a single dose not exceeding 800 mg; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Cisplatin Injection: Administration and Dosage: Intravenous infusion, 75 mg/m^2; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Interventions: Drug: BEBT-109 Capsules; Drug: Pemetrexed Disodium for Injection; Drug: Carboplatin Injection; Drug: Cisplatin Injection
- BEBT-109 monotherapy (Experimental): BEBT-109 Capsules: Administration and Dosage: Oral administration, 180mg; Frequency and Duration of Administration: Once a day,and 21 days as a treatment cycle.
  Interventions: Drug: BEBT-109 Capsules

INTERVENTIONS:
Drug: BEBT-109 Capsules — BEBT-109 Capsules: Administration and Dosage: Oral administration, 120mg or 180mg; Frequency and Duration of Administration: Once a day or twice a day,and 21 days as a treatment cycle.
  Other Names: KCBT-1083
Drug: Pemetrexed Disodium for Injection — Pemetrexed Disodium for Injection: Administration and Dosage: Intravenous infusion, 500mg/m^2; Frequency and Duration of Administration: On the first day of each cycle,and 21 days as a treatment cycle.
  Arms: Dose group A of BEBT-109 combined with investigator-selected chemotherapy; Dose group B of BEBT-109 combined with investigator-selected chemotherapy; Dose group C of BEBT-109 combined with investigator-selected chemotherapy
Drug: Carboplatin Injection — Carboplatin Injection: Administration and Dosage: Intravenous infusion, AUC=5 mg/ml.min, with a single dose not exceeding 800 mg; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Arms: Dose group A of BEBT-109 combined with investigator-selected chemotherapy; Dose group B of BEBT-109 combined with investigator-selected chemotherapy; Dose group C of BEBT-109 combined with investigator-selected chemotherapy
Drug: Cisplatin Injection — Cisplatin Injection: Administration and Dosage: Intravenous infusion, 75 mg/m^2; Frequency and Duration of Administration: On the first day of each cycle for the first four cycles, and 21 days as a treatment cycle, totaling four cycles.
  Arms: Dose group A of BEBT-109 combined with investigator-selected chemotherapy; Dose group B of BEBT-109 combined with investigator-selected chemotherapy; Dose group C of BEBT-109 combined with investigator-selected chemotherapy

SUMMARY:
This is a multicenter, open Phase II clinical study to evaluate the efficacy, safety, and pharmacokinetic characteristics of BEBT-109 combined with injectable pemetrexed disodium and carboplatin or cisplatin injection as first-line treatment for locally advanced, recurrent, or metastatic non-small cell lung cancer carrying EGFR exon 20 insertion mutations.

DETAILED DESCRIPTION:
This study initially sets up two cohorts. In cohort 1, the treatment is BEBT-109 combined with investigator-selected chemotherapy (injectable pemetrexed disodium combined with carboplatin or cisplatin injection). In cohort 2, the treatment is BEBT-109 monotherapy (BEBT-109 capsule at a dose of 180mg, taken orally once daily). Based on different dosing regimens of BEBT-109 capsules, cohort 1 is divided into three dose groups: A (BEBT-109 capsule at a dose of 180mg, taken orally once daily), B (BEBT-109 capsule at a dose of 120mg, taken orally twice daily), and C (BEBT-109 capsule at a dose of 120mg, taken orally once daily). Dose group A will first enroll six subjects to receive one cycle (a treatment cycle is 21 days) of drug treatment, and the safety data of subjects in dose group A will determine whether to adjust the dose for cohort 1 or to initiate other dose groups. If ≤2 subjects experience dose-limiting toxicity (DLT) during the DLT observation period, dose group A will be expanded to 20-30 subjects, and the decision to initiate dose group B will be made jointly by the investigators and the sponsor. If more than 2 subjects experience DLT, the decision to continue the study or to initiate dose group C will be made jointly by the investigators and the sponsor. Subjects in dose groups B and C will also initially enroll six subjects to undergo DLT safety follow-up, and then the decision to expand to 20-30 subjects will be made jointly by the investigators and the sponsor.

The decision to initiate cohort 2 will be based on the safety and efficacy results from cohort 1.

Each subject's study process includes three phases: screening, treatment, and follow-up. During the treatment period, subjects will undergo tumor assessments every 6 weeks ± 7 days. After discontinuing treatment, subjects will enter the follow-up period, where subjects without progressive disease (PD) will receive efficacy follow-up every 6 weeks ± 7 days (until tumor progression, death, or other antitumor treatment is initiated), and survival follow-up every 3 months (± 2 weeks). All subjects will receive study drug treatment until PD, death, intolerable toxicity occurs, or the subject withdraws informed consent (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Participants have a comprehensive understanding, voluntarily sign the Informed Consent Form (ICF), and are capable of completing all trial procedures;
2. Age ≥18 years old, both males and females are eligible;
3. According to the 8th edition of the American Joint Committee on Cancer（AJCC）TNM staging criteria for lung cancer: patients with histologically or cytologically confirmed non-squamous non-small cell lung cancer (NSCLC) that is unresectable and intolerant or refuses radical synchronous radiochemotherapy, with locally advanced (stage IIIB or IIIC), recurrent, or metastatic (stage IV) disease;
4. No prior systemic treatment for locally advanced (stage IIIB or IIIC) or recurrent/metastatic (stage IV) NSCLC. Note: 1) Neoadjuvant/adjuvant therapy is allowed as long as it has been completed at least 6 months before the disease is diagnosed as locally progressive or metastatic tumor; 2) Participants who have failed treatment with savolitinib in the past are allowed;
5. EGFR exon 20 insertion mutations confirmed by peripheral blood or tumor tissue testing conducted by a tertiary hospital or a qualified third-party testing agency, and records must be provided. Patients may have only EGFR exon 20 insertion mutations or may also have other EGFR or HER2 mutations;
6. At least one measurable lesion that meets the RECIST V1.1 criteria during the screening period. Lesions previously treated with radiotherapy cannot be used as target lesions unless there is clear radiological progression after radiotherapy;
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1, and no decline in performance status within two weeks before the screening period, with an expected survival time ≥12 weeks;
8. Provided that the subject has not received blood transfusion, erythropoietin, recombinant human thrombopoietin, or colony-stimulating factor treatment within 14 days before the screening period, laboratory tests indicate that the subject has adequate organ function, including:

   * Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥100×10^9/L; Hemoglobin (HGB) ≥90 g/L;
   * Total serum bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) (for patients with Gilbert's syndrome, total bilirubin ≤3×ULN is allowed);
   * AST and ALT ≤2.5×ULN (for those with liver metastasis, AST and ALT ≤5×ULN is allowed);
   * Creatinine clearance ≥45 ml/min (calculated according to the Cockcroft-Gault formula), and urine protein ≤1+ or for subjects with urine protein ≥2+, the 24-hour urine protein total is ≤1 g/24 h;
   * Activated partial thromboplastin time (APTT) ≤1.5×ULN, prothrombin time (PT) ≤1.5×ULN, international normalized ratio (INR) ≤1.5×ULN;
9. Participants with a history of liver cirrhosis have a Child-Pugh score of A or B ≤7 at screening;
10. The QT interval evaluated by ECG at screening is normal, defined as the corrected QT interval (Fridericia) (QTcF) ≤450 ms (for males) or ≤470 ms (for females) (those not meeting the standard need to be retested twice, and the average corrected value of the three measurements is taken);
11. Male and female participants of childbearing potential must agree to use reliable contraceptive methods (hormonal or barrier methods) during the study period and for at least 6 months after the last administration of the drug, and must not breastfeed, with a negative blood pregnancy test before the first administration.

Exclusion Criteria:

1. History of severe allergic diseases (such as uncontrollable asthma), severe drug (including investigational drugs not yet marketed) allergies, or known allergies or intolerance to any drug or drug component in this study;
2. Diagnosis of other primary malignant tumors besides NSCLC, except for the following: non-melanoma skin cancer or cervical carcinoma in situ that has been adequately treated and cured, non-metastatic prostate cancer, or other primary malignant tumors that have been clearly recurrence-free for at least 3 years since the last treatment and have a low potential risk of recurrence;
3. Major surgical procedures within 28 days before the first administration of the study drug, planned surgery during the study period, or postoperative complications from surgery performed within 2 months before the first administration of the study drug (except for minor surgeries that the investigator deems do not affect participation in the trial, such as catheter placement or minimally invasive biopsy);
4. Presence of pleural effusion, ascites, or pericardial effusion with significant symptoms or requiring drainage;
5. Poorly controlled diabetes mellitus. Definition: Hemoglobin A1C (HbA1c) ≥8%; or 7% ≤ Hemoglobin A1C < 8%, accompanied by clinical symptoms of diabetes, such as polyuria, polydipsia, polyphagia, and weight loss. (Subjects who have not been adequately treated to control blood sugar, after adjusting the drug treatment plan, with fasting blood glucose ≤10 mmol/L, and deemed suitable to participate in this study by the investigator, can be included);
6. Received live vaccines within 28 days before the first administration of the study drug or plan to receive any live vaccines during the study period;
7. Subjects with a tendency to bleed or evidence of bleeding, including:

   1. History of active ulcers or perforations of the stomach and duodenum within 6 months before the first dose, persistent positive fecal occult blood, history of gastrointestinal bleeding such as ulcerative colitis;
   2. History of hemoptysis (defined as blood that is bright red or 2.5 ml) within 2 weeks before the first dose, or the presence of unhealed wounds, ulcers, or fractures;
   3. Vasculitis;
   4. Other conditions that may cause bleeding as determined by the investigator;
8. Presence of severe gastrointestinal functional abnormalities that may affect the intake, transport, or absorption of the test drug (such as inability to swallow, uncontrollable vomiting, history of extensive gastrointestinal resection, chronic diarrhea, long-term use of proton pump inhibitors (PPIs) for gastric diseases, Crohn's disease, ulcerative colitis, intestinal obstruction, etc.);
9. Presence of central nervous system (CNS) metastasis, except for those who are asymptomatic, have stable disease, and do not require drug treatment within 4 weeks before the start of the study treatment;
10. Current spinal cord compression (symptomatic or asymptomatic, and detected by radiographic examination) or suspected meningeal disease (symptomatic or asymptomatic);
11. Imaging (CT or MRI) shows that the tumor invades major blood vessels or is not clearly demarcated from major blood vessels;
12. Significant clinical cardiovascular and cerebrovascular diseases within 6 months before the first study drug administration, including but not limited to:

    e. Acute myocardial infarction, unstable angina; f. New York Heart Association (NYHA) class III or IV congestive heart failure; g. Left ventricular ejection fraction <50% measured by echocardiography or multigated acquisition (MUGA) scan or with severe wall motion abnormalities; h. History of clinically significant ventricular arrhythmias (such as sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes); i. Subjects with poorly controlled hypertension, with systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg; j. Arterial/venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism; low molecular weight heparin treatment is allowed, and the use of nonsteroidal anti-inflammatory drugs (NSAIDs) or antiplatelet drugs (such as aspirin (>325 mg/day), clopidogrel (>75 mg/day), dipyridamole, ticlopidine, or cilostazol, etc.) is prohibited throughout the study period; k. Other arrhythmias deemed unsuitable for inclusion in this study by the investigator (such as third-degree atrioventricular block);
13. Presence of other severe or uncontrolled diseases that the investigator deems unsuitable for participation in this clinical trial or may affect the subject's compliance with the study protocol, including but not limited to:

    1. Interstitial lung disease, radiation pneumonitis or drug-related pneumonitis requiring steroid treatment;
    2. History of uncontrolled hereditary or acquired thrombotic diseases;
    3. Persistent or active infections, including but not limited to: hepatitis B virus (meeting both hepatitis B surface antigen positive or hepatitis B e antigen positive, and HBV-DNA greater than the upper limit of normal of the center's laboratory), hepatitis C virus (meeting both HCV-Ab positive and HCV-RNA positive), human immunodeficiency virus (HIV-Ab positive), syphilis non-specific antibody positive (rapid plasma reagin [RPR] or toluidine red unheated serum test [TRUST]) without clinical symptoms, or other active infections that require systemic treatment within 14 days before the first study drug administration;
    4. Severe or unhealed wounds, ulcers, or fractures;
14. History of drug or alcohol abuse or mental illness;
15. Use of drugs or herbal supplements that are strong inhibitors or inducers of CYP 3A4 and CYP 2C8 within 14 days before the first administration of the study drug ;
16. Received >30Gy of non-thoracic radical radiotherapy within 28 days before the first dose, >30Gy of thoracic radiotherapy within 24 weeks before the first dose, and ≤30Gy of palliative radiotherapy within 14 days before the first dose;
17. Participation in another clinical trial and drug administration within 4 weeks before the first dose;
18. Other conditions deemed unsuitable for entry into this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
ORR | Every 6 weeks,assessed up to 24 months.
  Objective response rate
AE | From the first administration of the study drug to 28 days after the last administration of the study drug.
  Adverse event

SECONDARY OUTCOMES:
DCR | Every 6 weeks,assessed up to 24 months.
  Disease control rate

OTHER OUTCOMES:
DOR | Every 6 weeks,assessed up to 24 months.
  Duration of response
PFS | Every 6 weeks,assessed up to 24 months.
  Progression-free survival
OS | From date of administration until date of death from any cause, assessed up to 24 months.
  Overall survival
TTR | Every 6 weeks,assessed up to 24 months.
  Time to response
Tmax | From 1 hour before dosing on day 1 and day 20 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 18 and day 19 of the first cycle (each cycle is 21 days).
  Time of peak plasma concentration
Cmax | From 1 hour before dosing on day 1 and day 20 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 18 and day 19 of the first cycle (each cycle is 21 days).
  Peak plasma concentration
t1/2 | From 1 hour before dosing on day 1 and day 20 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 18 and day 19 of the first cycle (each cycle is 21 days).
  Half-life of plasma drug concentrations
AUC0-t | From 1 hour before dosing on day 1 and day 20 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 18 and day 19 of the first cycle (each cycle is 21 days).
  Area under the plasma concentration time curve from 0 hour to last time of quantifiable concentration after administration
CL | From 1 hour before dosing on day 1 and day 20 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 18 and day 19 of the first cycle (each cycle is 21 days).
  Apparent plasma clearance

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China